CLINICAL TRIAL: NCT05588583
Title: A Prospective, Open, Multi-Center, Interventional, Non-Comparative Clinical Investigation to Follow the Progress of Exuding Chronic Wounds Using Mepilex® Up
Brief Title: A Clinical Investigation to Follow the Progress of Exuding Chronic Wounds Using Mepilex® Up as the Primary Dressing.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DIPLO01
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2022-10

CONDITIONS: Wounds; Wound of Skin; Wound Leg; Wound; Foot; Diabetic Foot Ulcer; Venous Leg Ulcer
Keywords: Diabetic Foot Ulcer; Venous Leg Ulcer
MeSH Terms: conditions — Wounds and Injuries; Foot Injuries; Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: The model is a prospective, open, multi-center, interventional, non-comparative investigation with the aim to follow exuding chronic wound progression for 6 weeks according to local standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Supportive Care with Mepilex Up (Experimental): All Subjects will use a soft, silicone, non-bordered, adhesive, foam dressing called Mepilex Up as the absorbent primary dressing.
  Interventions: Device: Mepilex Up

INTERVENTIONS:
Device: Mepilex Up — Mepilex Up is a highly conformable dressing that absorbs both low and high viscous exudates, maintains a moist wound environment and minimises the risk of maceration. The dressing has a Safetac® wound contact layer that is a unique adhesive technology. It minimises pain to patients and trauma to wounds and the surrounding skin at dressing removal.
  Mepilex Up consists of:
  * a soft silicone wound contact layer (Safetac)
  * a flexible absorbent pad of compressed polyurethane foam
  * an outer polyurethane film which is breathable but waterproof
  Dressing material content:
  Silicone, polyurethane

SUMMARY:
The goal of this clinical trial is to follow the progress of wounds in those with venous leg ulcers and diabetic foot ulcers while using an absorbent dressing called Mepilex Up. The main objective is to follow the progress of these wounds over time from initial visit to each follow-up visit.

Participants will be asked to wear Mepilex Up dressing for up to 6 weeks of treatment or until healed, changed at every one-week interval.

DETAILED DESCRIPTION:
This investigation is designed as a prospective, open, multi-center, interventional, non-comparative investigation with the aim to follow exuding chronic wound progression for 6 weeks according to local standard of care. Wound progress is a summary endpoint of the total effect of treatment using Mepilex Up as the absorbent dressing and includes the changes in an objectively measured wound area and subjectively evaluated wound condition. Two indications will be included: Venous Leg Ulcers (VLU) and Diabetic Foot Ulcers (DFU). A total of n=68 participants, approximately 34 per indication, will be recruited at up to 8 centers in the US.

There will be a total of seven (7) visits to the investigation site for participants during the treatment period: baseline, followed by weekly visits up to six (6) weeks post baseline. During visits, evaluations will be performed to assess wound progression and status, wound dressing properties, as well as Subject pain, comfort, and quality of life. Safety will be assessed at all visits. One target wound per participant will be included in this investigation.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent to participate (including consent for digital imaging)
* Adult aged ≥18 years
* Diagnosed with a chronic, exuding VLU or DFU
* Exudate amount moderate to large
* Wound size from 3 cm2 to 30 cm2 for VLU and ≥1 cm2 for DFU, as determined by the clinician
* For VLU: ABPI (within 3 months) > 0.7. If ABPI > 1.4, then big toe pressure > 60 mmHg is required or an alternative measurement verifying normal distal arterial flow
* For VLU: Willing to be compliant with compression therapy

Exclusion Criteria:

* Infected ulcer according to the judgment of the investigator defined as any wound condition requiring the prescription or continuation of systemic antibiotic therapy at enrollment
* Circumferential wound
* Known allergy/hypersensitivity to the materials of the dressing
* Patients participating in the DIPLO NBF study
* Use of wound fillers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Wound progress of the total effect of treatment using Mepilex Up | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  Wound progress is the total effect of treatment using Mepilex Up as the absorbent dressing and includes the changes in an objectively measured wound area and subjectively evaluated wound condition by the treating investigator/designee. Wound progress will be assessed as deteriorated, no change, improved, or healed at each visit. Wound area will be measured by an independent evaluator assisted by digital software at each visit and recorded as cm2 using the formula, A= π*L*W/4.

SECONDARY OUTCOMES:
Percentage wound area reduction over time | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  The percentage of wound area (cm2) reduction over time will be assessed by a formula as the area of an ellipse and measured by an independent evaluator assisted by digital software on all digital photographs taken at each scheduled visit.
Percentage wound volume reduction over time (DFUs only) | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  The percentage wound volume (cm3) reduction over time will be calculated by a formula from the manually assessed wound depth and the digitally assessed wound area.
Linear wound healing over time | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  The linear wound healing will be calculated with Gilman's formula (cm/day), G = - (A1-A0)/ {[(P1+P0)/2]*(t1-t0)}, where:
  A0 = previous visit area A1 = current visit area P0 = previous visit perimeter P1 = current visit perimeter t0 = previous visit time t1 = current visit time.
  Area (A) and Perimeter (P) will be assessed by an independent evaluator assisted by digital software. Perimeter (P) will be measured in cm and Area (A) will be assessed in cm2.
Change in granulation tissue over time | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  The area of wound covered by granulation tissue, (%) before and after cleansing/debridement will be assessed as follows: 1) via an independent evaluator assisted by digital software; and 2) via visual judgement by investigator/designee and determined as: None, 1%-24%, 25%-49%, 50%-74%, or 75%-100%.
Change in sloughy tissue over time | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  The area of wound covered by sloughy tissue, (%) before and after cleansing/debridement will be assessed as follows: 1) via an independent evaluator assisted by digital software; and 2) via visual judgement by investigator/designee and determined as: None, 1%-24%, 25%-49%, 50%-74%, or 75%-100%.
Change in exudate amount over time | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  Exudate amount will be captured as a subjective measure from the investigator/designee and assessed as none, scant, small, moderate, or large.
Change in exudate nature over time | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  Exudate nature will be captured as a subjective measure from the investigator/designee via the following category descriptive scale: serous, serosanguinous, sanguineous, seropurulent, fibrinous, purulent, hemopurulent, or hemorrhagic.
Change in peri-wound skin condition over time | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  The change in peri-wound skin condition over time will be assessed by visual assessment (No/Yes) by investigator/designee for maceration, dry skin, erythema/redness, and other peri-wound skin conditions. The Transepidermal Water Loss, or TEWL, will be an additional variable assessed at every visit for VLU Subjects at a limited number of clinical sites. TEWL measurements will be done using a portable VapoMeter.
Change in maceration over time | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  Area of wound covered by macerated tissue (%) will be assessed before debridement in cm2 by an independent evaluator assisted by digital software.
  The maximal distance (cm) from as close to the wound edge as possible to the end of maceration, assessed from wound photo, taken before debridement, by an independent evaluator assisted by digital software. The area of maceration will be assessed from a wound photo taken before debridement by an independent evaluator assisted by digital software.
Wound/Peri-Wound itch score prior to dressing removal over time (PRO) | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  The Subject itch severity before dressing removal over time will be assessed at all follow-up visits using the Numerical Rating Scale (NRS). The Subject verbally rates their level of itchiness on a level from 0 to 10, where 0 indicates no itch and 10 is the worst itch.
Wound pain score during dressing wear over time (PRO) | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  Subject pain severity during dressing wear over time will be assessed at all follow-up visits using the Numerical Rating Scale (NRS). The Subject verbally rates the pain on a level from 0 to 10, where 0 indicates no pain and 10 is the worst pain.
Wound pain score related to removal of dressing over time (PRO) | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  Subject pain severity at dressing removal will be assessed at all follow-up visits using the NRS scale where the Subject verbally rates the pain on a level from 0 to 10, where 0 indicates no pain and 10 is the worst pain. Any pre-procedural or intra-procedural pain medication administered at the time of dressing removal will be recorded.
Trauma to the wound/peri-wound during dressing removal over time | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  Trauma to the wound will be captured via visual judgement by the investigator/desginee using an ordinal scale of none, very slight, moderate, or high. Trauma to the peri-wound skin will be captured via visual judgement by the investigator/designee using the ordinal scale of none, very slight, moderate, or high.
Primary dressing's ability to be comfortable to wear (PRO) | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  Subjects will be asked to rate Mepilex Up degree of comfort using a 4-item scale of very poor, poor, good, or very good.
For VLU: Mepilex Up ability to be comfortable to wear with compression (PRO) | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  VLU Subjects will be asked to rate Mepilex Up degree of comfort while wearing with compression using a 4-item scale of very poor, poor, good, or very good.
For DFU: Mepilex Up ability to be comfortable to wear with offloading (PRO) | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  DFU Subjects will be asked to rate Mepilex Up degree of comfort while wearing with offloading using a 4-item scale of very poor, poor, good, or very good.
Evaluation of Wound Quality of Life (QoL) (PRO) | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  A Wound-QoL-17 questionnaire will be completed by each Subject to measure the disease-specific, health-related QoL of those with chronic wounds. All items assess impairments within the preceding seven days.
Technical Performance (Investigator/designee's evaluation) | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  Several questions will be asked to evaluate the technical performance properties of Mepilex Up. The following will be assessed by the investigator/designee using no/yes values: 1) Occurrence of strike-through, defined as the inability of the dressing to stay sealed over the wound causing leakage of wound exudate; and 2) Occurrence of product residue in the wound bed or on peri-wound skin after dressing removal. All other properties will be assessed by the investigator/designee using a 4-item scale of very poor, poor, good, very good. These include:
  * Ability to absorb exudates with different viscosities,
  * Ability to retain exudate,
  * Ease of application,
  * Ability to conform to the wound during wear,
  * Ability to be repositioned during application,
  * Inability to adhere to moist wound bed,
  * Ability to adhere to healthy, intact skin,
  * Ability to stay on during application and use,
  * Overall satisfaction with the dressing's properties.
Status of dressing during a routine dressing change or complication | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  The status of Mepilex Up during a routine dressing change or complication will be assessed by the investigator/designee as strike-through, saturated, displaced/slipping, or other. This will be recorded in the Dressing Log.
Pre-compression edema | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  The specification of any pre-compression edema prior to applying/changing compression therapy will be assessed by the investigator/designee as:
  * 0 (no clinical edema)
  * 1+ (≤2 mm indentation)
  * 2+ (2-4 mm indentation)
  * 3+ (4-6 mm indentation)
  * 4+ (6-8 mm indentation)
Compression removed/changed/applied | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  Assessment of compression by the investigator/designee will cover:
  * Compression removal (No/Yes)
  * Compression changed/applied (No/Yes)
  * Type of compression used
Compliance with compression | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  The investigator/designee will evaluate Subject compliance with compression. Assessment will include being fully compliant (defined as 7 out of 7 days with compression), moderately compliant (defined as 1 to 3 days without compression out of 7 days), or not compliant (defined as >3 days without compression out of 7 days).
Offloading Use/Type | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  The assessment of offloading will cover if it were used (No/Yes) and specification of offloading type by the investigator/designee.
Compliance to offloading | A maximum total treatment period of 44 days or until healed, whichever occurs first.
  The investigator/designee will evaluate Subject compliance with offloading. Assessment will include being fully compliant (defined as 7 out of 7 days with offloading), moderately compliant (defined as 1 to 3 days without offloading out of 7 days), or not compliant (defined as >3 days without offloading out of 7 days).
Wear time (days) | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  Wear time will be determined from the Subject Dressing Log at each visit by collecting:
  * Date of dressing application/change
  * Reason for change application/change
  * Lot/batch
  * Size
  * Quantity
Debridement performed | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  The following debridement details will be recorded for each Subject at each visit:
  * Debridement performed (No/Yes)
  * Debridement method
  * Ease of debridement (Very easy/Easy/Difficult/Very Difficult)
Cleansing performed | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  The following cleansing details will be recorded for each Subject at each visit:
  * Cleansing performed (No/Yes)
  * Type of cleansing agent used
Evaluation of all reported adverse events and device deficiencies | From baseline visit to last follow-up visit, a maximum total treatment period of 44 days or until healed, whichever occurs first.
  If any reported adverse events or device deficiencies are reported, an evaluation will take place to determine root cause.

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, MAS, Principal Investigator — University of Miami
Locations (4):
- United States (4):
  - Center for Clinical Research, Inc., Castro Valley, California
  - Felix Sigal, DPM, Los Angeles, California
  - University of Miami, Miami, Florida
  - Serena Group Research Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gould L, Abadir P, Brem H, Carter M, Conner-Kerr T, Davidson J, DiPietro L, Falanga V, Fife C, Gardner S, Grice E, Harmon J, Hazzard WR, High KP, Houghton P, Jacobson N, Kirsner RS, Kovacs EJ, Margolis D, McFarland Horne F, Reed MJ, Sullivan DH, Thom S, Tomic-Canic M, Walston J, Whitney J, Williams J, Zieman S, Schmader K. Chronic wound repair and healing in older adults: current status and future research. Wound Repair Regen. 2015 Jan-Feb;23(1):1-13. doi: 10.1111/wrr.12245. Epub 2015 Feb 13. PMID 25486905
- [Background] Tickle J. Wound exudate: a survey of current understanding and clinical competency. Br J Nurs. 2016 Jan 28-Feb 10;25(2):102-9. doi: 10.12968/bjon.2016.25.2.102. PMID 27119542
- [Background] Gonzalez de la Torre H, Quintana-Lorenzo ML, Perdomo-Perez E, Verdu J. Correlation between health-related quality of life and venous leg ulcer's severity and characteristics: a cross-sectional study. Int Wound J. 2017 Apr;14(2):360-368. doi: 10.1111/iwj.12610. Epub 2016 Apr 25. PMID 27112627
- [Background] Jones JE, Robinson J, Barr W, Carlisle C. Impact of exudate and odour from chronic venous leg ulceration. Nurs Stand. 2008 Jul 16-22;22(45):53-4, 56, 58 passim. doi: 10.7748/ns2008.07.22.45.53.c6592. PMID 18686695
- [Background] Maume S, Van De Looverbosch D, Heyman H, Romanelli M, Ciangherotti A, Charpin S. A study to compare a new self-adherent soft silicone dressing with a self-adherent polymer dressing in stage II pressure ulcers. Ostomy Wound Manage. 2003 Sep;49(9):44-51. PMID 14581709
- [Background] Moore Z, Strapp H. Managing the problem of excess exudate. Br J Nurs. 2015 Aug 13-Sep 19;24(15):S12, S14-7. doi: 10.12968/bjon.2015.24.Sup15.S12. PMID 26266558
- [Background] Rippon M, Davies P, White R. Taking the trauma out of wound care: the importance of undisturbed healing. J Wound Care. 2012 Aug;21(8):359-60, 362, 364-8. doi: 10.12968/jowc.2012.21.8.359. PMID 22885308
- [Background] Gorin DR, Cordts PR, LaMorte WW, Manzoian JO. The influence of wound geometry on the measurement of wound healing rates in clinical trials. J Vasc Surg. 1996 Mar;23(3):524-8. doi: 10.1016/s0741-5214(96)80021-8. PMID 8601898
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Augustin M, Conde Montero E, Zander N, Baade K, Herberger K, Debus ES, Diener H, Neubert T, Blome C. Validity and feasibility of the wound-QoL questionnaire on health-related quality of life in chronic wounds. Wound Repair Regen. 2017 Sep;25(5):852-857. doi: 10.1111/wrr.12583. Epub 2017 Nov 2. PMID 29080332
- [Background] Rippon M WM, Bielfeldt S. An evaluation of properties related to wear time of four dressings during a five-day period. Wounds UK. 2015;11(1):45-54.
- [Background] Young T, Clark M, Augustin M, Carville K, Curran J, Flour M, et al. International consensus. Optimising wellbeing in people living with a wound. An expert working group review. Wounds International; London 2012.
- [Background] Chadwick P, McCardle J. Exudate management using a gelling fibre dressing. The Diabetic Foot Journal. 2015;18(1):43-8.
- [Background] World Union of Wound Healing Societies (WUWHS). Principles of best practice: Wound exudate and the role of dressings. A consensus document. 2019.
- [Background] European Wound Management Association (EWMA). Position document: Wound bed preparation in practice. London: MEP Ltd. 2004.
- [Background] Romanelli M, Vowden K, Weir D. Exudate Management Made Easy Wounds International 2010.
- [Background] Walker M, Parsons D. Hydrofiber® technology: its role in exudate management. Wounds UK; 2010. p. 31-38.
- [Background] Fletcher J. Development of a new wound assessment form, Clinical practice development. Wounds UK. 2010;6(1).